CLINICAL TRIAL: NCT05482451
Title: Treatment With Nivolumab and All-trans Retinoic Acid for Patients With Refractory Pancreatic Cancer
Brief Title: Nivolumab and All-trans Retinoic Acid for Pancreatic Cancer
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMUH110-REC1-013
Record Dates: First submitted 2022-07-27; First posted 2022-08-01 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Effect of Drug
Keywords: Pancreatic cancer; Nivolumab; All-trans retinoic acid; Vesanoid; ADAR1
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Nivolumab; Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab + all-trans retinoic acid (Experimental): Nivolumab: 3mg/kg intravenously on day 1.
  All-trans retinoic acid (Vesanoid) 45 mg/m2 on days 1-14. The dose of Vesanoid can be increased with addition of 15 mg/m2 in next course of treatment if there is no severe adverse effects. Therefore, the dose of Vesanoid could be 60 mg/m2 from the second course, 75 mg/m2 from the third course, till the maximal dose of 150 mg/m2 if patients tolerated the treatment. The decision of dose escalation is left to in-charge physician.
  The treatment cycle will repeat every 2 weeks.
  Interventions: Drug: Nivolumab; Drug: all trans retinoic acid

INTERVENTIONS:
Drug: Nivolumab — Nivolumab, an immune checkpoint inhibitors targeting PD-1, represents a popular treatment option for patients with cancers via immunological mechanism. However, previous studies using nivolumab alone in pancreatic cancer have failed.
  Other Names: Opdivo
Drug: all trans retinoic acid — Our previous basic studies revealed that all-trans retinoic acid repressed pancreatic adenocarcinoma cell growth and colony formation. All-trans retinoic acid represses ADAR1, a member of interferon-stimulated genes and a negative regulator of IFNs signaling. On the other hand, all-trans retinoic acid simultaneously increases PD-L1 expression for cancer cells to evade immune surveillance. Since combination of anti-PD1 antibody and all-trans retinoic acid may block self-regulating negative feedback loops of IFNs response, this therapeutic strategy may improve outcomes of pancreatic adenocarcinoma patients.
  Other Names: Vesanoid

SUMMARY:
This study is to examine the anticancer activity of the combination therapy with all-trans retinoic acid and nivolumab in patients with chemotherapy-refractory advanced or metastatic pancreatic adenocarcinoma.

DETAILED DESCRIPTION:
Pancreatic cancer is an aggressive and lethal disease. Even two combination regimens, FOLFIRINOX and albumin-bound paclitaxel in combination with gemcitabine, are superior to gemcitabine alone as the first-line treatments, the prognosis of patients with locally advanced or metastatic pancreatic cancer remains poor, with a median overall survival of 8 to 11 months and an estimated 2-year survival of only 2%. Even more, there is currently no available treatment proven beneficial for patients who fail the second-line therapy with liposomal irinotecan in combination with 5-FU.

Immune checkpoint inhibitors targeting PD-1 or PD-L1 represent a popular treatment option for patients with some kinds of cancers, but previous studies in pancreatic cancer have failed. One critical challenge for immunotherapy in pancreatic cancer is to find efficient therapeutic approaches to reverse this "cold" tumor into a "hot" tumor. Our previous basic studies revealed that all-trans retinoic acid repressed pancreatic adenocarcinoma cell growth and colony formation. Set-to-set genetic analysis revealed that genes regulated by all-trans retinoic acid were predominantly involved in immune response including interleukin-6, tumor necrotic factor-α, IFNs signaling, and PD-L1. Furthermore, mice bearing pancreatic cancer treated with combination of anti-PD-1 and all-trans retinoic acid had a significantly longer survival compared to mice treated with anti-PD-1 or all-trans retinoic acid alone.

Based on the previous findings, we propose this pilot, compassionate use of combination therapy with all-trans retinoic acid and nivolumab for patients with locally advanced or metastatic pancreatic adenocarcinoma who are refractory to current available treatment. This study will also examine ADAR1 as a novel prognostic and predictive biomarker for pancreatic adenocarcinoma patients. This study will help to delineate the role of ADAR1 as a predictive biomarker for immunotherapy, all-trans retinoic acid as a suppressor of ADAR1, and most importantly, the combination of all-trans retinoic acid and nivolumab as an effective anticancer therapy for patients with pancreatic adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

Patients will be included in the study if they meet all of the following criteria:

1. Patients with age ≥ 20 years old
2. Histologically confirmed pancreatic adenocarcinoma
3. Unresectable locally advanced, recurrent or metastatic diseases ineligible or unsuitable for further surgical or radiation interventions
4. Documented disease progression within 6 months after standard chemotherapies or no available standard chemotherapy. The standard chemotherapies include gemcitabine, nab-paclitaxel, S-1, and FOLFIRINOX. Patient who has prior anti-PD1/anti-PD-L1 treatment will not be eligible.
5. ECOG Performance Status 0-2
6. Documented measurable disease as defined by RECIST v1.1
7. Adequate hematologic parameters, and hepatic and renal functions defined as

   1. absolute neutrophil count ≥ 1,000/μL
   2. platelets ≥ 75,000/μL
   3. total bilirubin ≤ 2.5X ULN (≤ 5X ULN if attributable to liver metastases)
   4. AST/ALT ≤ 2.5X ULN (≤ 5X ULN if attributable to liver metastases)
   5. serum creatinine ≤ 2 mg/dL or creatinine clearance ≥ 30 mL/min (by calculated or 24-hour urine collection)
8. Normal ECG or ECG without any clinical significant findings
9. Able to understand and sign an informed consent (or have a legal representative who is able to do so)

Exclusion Criteria:

Patients will be excluded from the study if they meet any of the following criteria:

1. History of allergic reaction to all-trans retinoic acid or nivolumab
2. Patient with liver cirrhosis with Child-Pugh score ≥ 8 (Late Child-Pugh B and Child-Pugh C)
3. Active CNS metastasis defined by clinical symptoms, cerebral edema, steroid or anti-convulsant requirement, or progressive growth. Patients with a history of CNS metastasis or cord compression are allowed in the study if they have been treated and are clinically stable
4. With clinically significant gastrointestinal disorder including bleeding, inflammation, occlusion or diarrhea > grade 1
5. With uncontrolled intercurrent illness that could limit study compliance or judged to be ineligible for the study by the investigators including, but not limited to, any of the following:

   1. ongoing or active infection requiring antibiotic treatment
   2. symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia
   3. psychiatric illness or social situation that would preclude study compliance
6. Pregnant or breast feeding women (a urine pregnancy test must be performed on all patients who are of childbearing potential before entering the study, and the result must be negative)
7. Patients taking the following medications: immunosuppressants, corticosteroids with the exception of administration topically (e.g., external, intra-articular, intranasal, ophthalmic, or inhalational use) or temporarily (e.g., for treatment or prophylaxis of contrast medium allergy or adverse events), antitumor therapies (e.g., chemotherapies, molecular-targeted therapies, immunotherapies), radiopharmaceuticals with the exception of diagnostic purposes, transplant therapies, vitamin A, antifibrinolytic agents (tranexamic acid, aminocaproic acid, aprotinin), inducers (rifampicin, glucocorticoids, phenobarbital and pentobarbital) or inhibitors (ketoconazole, cimetidine, erythromycin, verapamil, diltiazem and cyclosporine) of the hepatic P450 system, and other unapproved drugs (e.g., investigational use of drugs, unapproved combined formulations, unapproved dosage forms).

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Overall response | From the date of registration until the end of treatment, up to 2 years.
  Overall response is evaluated using Response Evaluation Criteria in Solid Tumors criteria (RECIST 1.1). A participant is considered to have responded if either of the following outcomes is achieved:
  1. Complete Response: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm
  2. Partial Response: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.

SECONDARY OUTCOMES:
Progression-free survival | From the date of registration until disease progression or death, up to 3 years.
  The median duration of time from the time of registration until disease progression or death. Disease progression is assessed using RECIST 1.1 criteria.

OTHER OUTCOMES:
Overall survival | From the date of registration to the date of patients death, up to 3 years.
  The median duration of time from the time of registration until death

CONTACTS AND LOCATIONS:
Overall Officials: Li-Yuan Bai, Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Please Select, Taiwan

IPD SHARING:
Plan to Share IPD: No
Age, basic informations

DOCUMENTS (1):
  • Study Protocol (2022-10-07): https://cdn.clinicaltrials.gov/large-docs/51/NCT05482451/Prot_000.pdf